CLINICAL TRIAL: NCT02857764
Title: SGLT2 Inhibitor Risk of Below-Knee Lower Extremity Amputation: A Retrospective Cohort Study Using a Large Claims Database in the United States
Brief Title: Sodium-glucose Co-transporter 2 (SGLT2) Inhibitor Risk of Below-Knee Lower Extremity Amputation: A Retrospective Cohort Study Using a Large Claims Database in the United States
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: RRA-17578; RRA-17578 (Other: Janssen Research & Development, LLC.)
Record Dates: First submitted 2016-08-03; First posted 2016-08-05 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Sodium-glucose Co-transporter 2 Inhibitors (SGLT2i) New Users: Participants will not receive any intervention as a part of this study. SGLT2i includes canagliflozin, dapagliflozin, empagliflozin as prescribed in clinical practice. Participants will be evaluated in 2 sub-cohorts (with or without high CV risk) and overall.
- Canagliflozin New Users: Participants will not receive any intervention as a part of this study. This cohort contains new users of canagliflozin as prescribed in clinical practice. Participants will be evaluated in 2 risk) and overall.
- Dapagliflozin New Users: Participants will not receive any intervention as a part of this study. This cohort contains new users of dapagliflozin as prescribed in clinical practice. Participants will be evaluated in 2 sub-cohorts (with or without high CV risk) and overall.
- Empagliflozin New Users: Participants will not receive any intervention as a part of this study. This cohort contains new users of empagliflozin as prescribed in clinical practice. Participants will be evaluated in 2 sub-cohorts (with or without high CV risk) and overall.
- First-time Non-SGLT2i AHA New Users: Participants will not receive any intervention as a part of this study. Non-SGLT2i AHA include dipeptidyl peptidase-4 (DPP-4) inhibitors, glucagon-like peptide-1 (GLP-1) agonists, thiazolidinediones (TZDs), Sulfonylureas, Insulin, and other AHAs. Participants will be evaluated in 2 sub-cohorts (with or without high CV risk) and overall.

SUMMARY:
The purpose of the study is to estimate the incidence of below-knee lower extremity amputation in type 2 diabetes mellitus (T2DM) participants newly exposed to sodium-glucose co-transporter 2 inhibitors (SGLT2i)/ non-SGLT2i antihyperglycemic agents (AHA) overall and in the subgroup with high cardiovascular (CV) risk and to compare the hazards of below-knee lower extremity amputation in canagliflozin new users versus non-SGLT2i AHA new users.

ELIGIBILITY:
Inclusion Criteria:

* First exposure to the particular drug in person's history
* For the initial analysis, exposure start is between April 1, 2013 and January 31, 2015. For the ongoing repeat analysis per the protocol amendment, the study period ending date will vary depending on the time of each data extraction and analysis
* At least 365 days of observation time prior to index
* At least 1 condition occurrence of 'Type II diabetes' any time before or on index
* Exactly 0 condition occurrences of 'Type I diabetes' any time before or on index

Exclusion Criteria:

* Participants who had amputations prior to the index date were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who are new users (with at least 365 day of prior observation) to a drug exposure of interest between April 1, 2013 and January 31, 2015 and at least 1 condition occurrence of 'Type II diabetes' any time before or on index and no condition occurrences of 'Type I diabetes' or 'Secondary diabetes' any time before or on index date. January 31, 2015 reflects the data cutoff date for the initial analysis.
Sampling Method: Non-Probability Sample
Enrollment: 127690 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Below-knee Lower Extremity Amputation in Type 2 Diabetes Mellitus (T2DM) Patients Newly Exposed to Sodium-glucose Co-transporter 2 Inhibitors (SGLT2i) Overall and in the Subgroup With High Cardiovascular (CV) Risk | up to 6 years (estimated study duration)
  The occurrence of a below-knee lower extremity amputation will be defined by observing an associated procedure code in the outpatient or inpatient medical service claims.
Incidence of Below-Knee Lower Extremity Amputation in T2DM Patients Newly Exposed To non-SGLT2i Aha Overall And In The Subgroup With High CV Risk | up to 6 years (estimated study duration)
  The occurrence of a below-knee lower extremity amputation will be defined by observing an associated procedure code in the outpatient or inpatient medical service claims.
Incidence of Below-Knee Lower Extremity Amputation in Canagliflozin New Users Versus non-SGLT2i Aha New Users | up to 6 years (estimated study duration)
  Hazard ratio will be estimated using a conditional Cox proportional hazards model based on propensity-matched cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC